CLINICAL TRIAL: NCT01846429
Title: A Phase I/II Study of Oral Bicarbonate as Adjuvant for Pain Reduction in Patients With Tumor Related Pain
Brief Title: Oral Bicarbonate as Adjuvant for Pain Reduction in Patients With Tumor Related Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs unavailable. Study did not progress to Phase 2.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Reliable Cancer Therapies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-17136
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Tumor; Cancer; Pain; Malignant Solid Tumor; Unresectable Malignant Neoplasm; Hematologic Malignancy; Multiple Myeloma; Lymphoma; Neoplasm Metastasis
Keywords: cancer; pain fibers; acid levels; tumor related pain; cancer related pain; sodium bicarbonate; pain reliever; metastatic; unresectable; solid malignancy; hematologic malignancy; multiple myeloma; lymphoma
MeSH Terms: conditions — Neoplasms; Pain; Hematologic Neoplasms; Multiple Myeloma; Lymphoma; Neoplasm Metastasis; Cancer Pain | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Bicarbonate Treatment (Experimental): A 3+3 design for Phase I component and a two staged design for Phase II were to be used. Treatment: Sodium Bicarbonate Capsules (900 mg).
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — Cohort 1 patients will take 10 capsules/day; cohort 2 patients will take 20 capsules/day; cohort 3 patients will take 30 capsules/day and cohort 4 patients will take 40 capsules/day. Cohort 2 - 4 patients will begin at the cohort 1 dose and dose escalate to their respective cohort doses in order to prevent any side effects associated with alkalosis. Dose escalation will occur at a rate of 10 capsules/week.

SUMMARY:
The purpose of this study is to:

* Determine how well people tolerate sodium bicarbonate taken by mouth in higher doses than those usually given for heartburn.
* Determine if sodium bicarbonate can reduce cancer-related pain.

DETAILED DESCRIPTION:
Single institution Phase I/II study of sodium bicarbonate in combination with standard medical management for patients with moderate to severe tumor related pain.

Patients with metastatic solid malignancies and patients with hematologic malignancies with moderate to severe tumor related pain on a stable opioid regimen will be the subjects of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic or unresectable solid malignancy or hematologic malignancy (multiple myeloma or lymphoma) and must have moderate to severe tumor related pain visual assessment scale (VAS)>4) on a stable or no opioid regimen (at least 3 days of an opiate regimen). VAS score should be greater than 4 at screening to be eligible.
* No planned palliative surgery, palliative radiotherapy for at least 4 weeks. However prior radiotherapy, and surgery is allowed and not limited to the number of procedures and courses. Concomitant chemotherapy with agents indicated in protocol guidelines (Tables 10 and 11B, Appendix IV) is allowed.
* No evidence of neurologic or psychiatric compromise which in the opinion of the investigator will interfere with completion of study assessments
* Age greater than 18 years and able to understand and sign the informed consent document
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status less than 3.
* A female patient and a male patient's female partner, of childbearing potential, must agree to use 2 adequate barrier methods of contraception to prevent pregnancy or to abstain from heterosexual activity throughout the study, starting from Visit 1, while receiving protocol-specified medication, and for 1 month after stopping the medication.

Exclusion Criteria:

* Patients with neuropathy and/or neuropathic pain as the only pain syndrome are not eligible.
* Patients with only chronic non-malignant pain are not eligible.
* Patients with renal insufficiency (creatinine > 2.5mg/dL) are excluded.
* Patients with history of congestive heart failure or pulmonary artery hypertension will be excluded.
* Patients with uncontrolled hypertension (systolic pressure >160, diastolic pressure >100) despite maximal antihypertensive therapy
* Patients unable to ingest sodium bicarbonate capsules (such as patients with dysphagia or severe nausea)
* Patients with ECOG performance status 3 or higher
* Patients with acute leukemia, myelodysplastic syndrome, and chronic myeloid leukemia are not eligible.
* Pregnant or lactating patients are not eligible.
* Patients with known allergy to sodium bicarbonate or patients with preexisting renal or acid base disorders for which sodium bicarbonate is contraindicated (such as metabolic alkalosis, severe congestive heart failure, hypernatremia, and hypocalcemia (see above))
* Patients with severe ongoing infections which places the patients at increased risks from therapy in the opinion of the investigator
* Patients receiving concomitant chemotherapy with agents indicated in protocol guidelines (Tables 10 and 11B, Appendix IV) or target therapy intended to prolong life within 2 weeks of starting the study drug
* Patients receiving experimental therapy within 2 weeks of starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Phase I - Maximum Tolerated Dose (MTD) | 4 weeks per participant
  To evaluate the safety (Phase I) of oral Sodium bicarbonate capsules as an adjuvant pain reliever in patients with tumor related moderate to severe pain.
  To determine the maximum tolerated dose (MTD) of oral sodium bicarbonate capsules for patients with tumor related moderate to severe pain.
Phase II - Percent of Participants With Desired Response | 4 weeks per participant
  Evaluate the efficacy (Phase II) of oral Sodium Bicarbonate capsules as an adjuvant pain reliever in patients with tumor related moderate to severe pain.
  Percent of patients with greater than 30% improvement in pain intensity by visual assessment scale at 4 weeks compared to baseline without a corresponding increase in opioid regimen. The response rate with 95% Clopper-Pearson confidence interval will be reported.

SECONDARY OUTCOMES:
Pain Measurement Ranking | 4 weeks per participant
  Pain will be rated by the participant using a visual assessment scale (VAS) on a 0 to 10 scale. Mild Pain (1-4), Moderate Pain (5-6), Severe Pain (7-10). The change in pain between baseline and 4 weeks after treatment as measured by the VAS will be assessed using two-sided one-sample t-test or Wilcoxon signed-rank test, depending on whether normality assumption holds.
Quality of Life (QOL) | 4 weeks per participant
  Quality of life will be assessed using the Memorial Symptom Assessment Scale (MSAS) and Brief Pain Inventory (BPI). The change in score between baseline and 4 weeks after treatment will be compared using two-sided one-sample t-test or Wilcoxon signed-rank test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mahipal, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Gillies RJ, Ibrahim-Hashim A, Ordway B, Gatenby RA. Back to basic: Trials and tribulations of alkalizing agents in cancer. Front Oncol. 2022 Nov 14;12:981718. doi: 10.3389/fonc.2022.981718. eCollection 2022. PMID 36452492